CLINICAL TRIAL: NCT00535405
Title: A Multicenter, Randomized, Double-Blind, Parallel, 12-Week Study to Evaluate the Efficacy and Safety of Ezetimibe/Simvastatin Combination Tablet Versus Atorvastatin in Elderly Patients With Hypercholesterolemia at High or Moderately High Risk for Coronary Heart Disease
Brief Title: A Study to Assess the Cholesterol Lowering Effect of Ezetimibe/Simvastatin Combination Tablet Compared to Another Cholesterol Lowering Drug in Elderly Patients With High Cholesterol at High or Moderately High Risk for Coronary Heart Disease (0653A-128)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Shering-Plough JV Study (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-128; 2007_588
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Results first posted 2010-05-25 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: High Cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): Each patient will receive 1 active treatment dose & 2 Placebo (Pbo) doses or 2 active treatment doses & 1 Pbo dose at randomization according to a predetermined partial blinding schedule to reduce the number of pills from 5 to 3 per patient per day for 12 weeks.
  Interventions: Drug: Atorvastatin 10 mg
- 2 (Experimental): Each patient will receive 1 active treatment dose & 2 Pbo doses or 2 active treatment doses & 1 Pbo dose at randomization according to a predetermined partial blinding schedule to reduce the number of pills from 5 to 3 per patient per day for 12 weeks.
  Interventions: Drug: Ezetimibe 10 mg/simvastatin 20 mg
- 3 (Experimental): Each patient will receive 1 active treatment dose & 2 Pbo doses or 2 active treatment doses & 1 Pbo dose at randomization according to a predetermined partial blinding schedule to reduce the number of pills from 5 to 3 per patient per day for 12 weeks.
  Interventions: Drug: Atorvastatin 20 mg
- 4 (Experimental): Each patient will receive 1 active treatment dose & 2 Pbo doses or 2 active treatment doses & 1 Pbo dose at randomization according to a predetermined partial blinding schedule to reduce the number of pills from 5 to 3 per patient per day for 12 weeks.
  Interventions: Drug: Ezetimibe 10 mg/simvastatin 40 mg
- 5 (Experimental): Each patient will receive 1 active treatment dose & 2 Pbo doses or 2 active treatment doses & 1 Pbo dose at randomization according to a predetermined partial blinding schedule to reduce the number of pills from 5 to 3 per patient per day for 12 weeks.
  Interventions: Drug: Atorvastatin 40 mg

INTERVENTIONS:
Drug: Atorvastatin 10 mg — Atorvastatin 10 mg and Placebo for ezetimibe and placebo for simvastatin once daily for 12 weeks
  Arms: 1
Drug: Ezetimibe 10 mg/simvastatin 20 mg — Ezetimibe 10 mg/simvastatin 20 mg and Placebo for atorvastatin once daily for 12 weeks
  Arms: 2
Drug: Atorvastatin 20 mg — Atorvastatin 20 mg and Placebo for ezetimibe and placebo for simvastatin once daily for 12 weeks
  Arms: 3
Drug: Ezetimibe 10 mg/simvastatin 40 mg — Ezetimibe 10 mg/simvastatin 40 mg and Placebo for atorvastatin once daily for 12 weeks
  Arms: 4
Drug: Atorvastatin 40 mg — Atorvastatin 40 mg and Placebo for ezetimibe and placebo for simvastatin once daily for 12 weeks
  Arms: 5

SUMMARY:
A multicenter study to evaluate the safety and efficacy of ezetimibe/simvastatin versus atorvastatin in elderly patients with high cholesterol at high or moderately high risk for coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a cholesterol level of 130 mg/dL or greater
* Patient is willing to maintain a cholesterol lowering diet for as long as they are in the study
* Patient is at moderate high risk or high risk for coronary heart disease per the National Cholesterol Education Program Adult Treatment Panel III (NCEP ATPIII) guidelines

Exclusion Criteria:

* Patient weighs less than 100 lbs
* Patient has an allergy to ezetimibe, simvastatin or atorvastatin

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1289 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Foody JM, Brown WV, Zieve F, Adewale AJ, Flaim D, Lowe RS, Jones-Burton C, Tershakovec AM. Safety and efficacy of ezetimibe/simvastatin combination versus atorvastatin alone in adults >/=65 years of age with hypercholesterolemia and with or at moderately high/high risk for coronary heart disease (the VYTELD study). Am J Cardiol. 2010 Nov 1;106(9):1255-63. doi: 10.1016/j.amjcard.2010.06.051. PMID 21029821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In 08-Nov-2007; Last Patient Last Visit 23-Mar-2009
  Eligible patients include drug-naïve patients or patients rendered naïve with the appropriate prior washout at moderately high or high risk for coronary heart disease 65 years and older.
Pre-assignment Details: The study evaluated patients ≥ 65 years of age at moderately high or high risk for Coronary Heart Disease (CHD), with or without atherosclerotic vascular disease. The study was a 3-week single-blind placebo run-in period and a 12-week active treatment period where patients were equally randomized to one of 5 treatment groups for 12 weeks
Groups:
- Atorvastatin 10 mg: Atorvastatin (Atorva) 10 mg once daily for 12 weeks
- Ezetimibe 10 mg/Simvastatin 20 mg: Ezetimibe (EZ) 10 mg/simvastatin (Simva) 20 mg once daily for 12 weeks
- Atorvastatin 20 mg: Atorvastatin 20 mg once daily for 12 weeks
- Ezetimibe 10 mg/Simvastatin 40 mg: Ezetimibe 10 mg/simvastatin 40 mg once daily for 12 weeks
- Atorva 40 mg: Atorvastatin 40 mg once daily for 12 weeks
Period: Overall Study
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg
Started | 257 | 259 | 259 | 257 | 257
Completed | 240 | 233 | 241 | 235 | 241
Not Completed | 17 | 26 | 18 | 22 | 16
Not completed — Adverse Event | 6 | 8 | 3 | 8 | 6
Not completed — Lost to Follow-up | 1 | 3 | 3 | 2 | 1
Not completed — Physician Decision | 3 | 2 | 0 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 11 | 10 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg | Total
Number analyzed (Participants) | 257 | 259 | 259 | 257 | 257 | 1289
Age, Continuous [Mean (Full Range); unit: years] | 72.1 [65 to 94] | 71.8 [65 to 95] | 71.7 [65 to 90] | 72.2 [65 to 96] | 72.1 [65 to 88] | 72.0 [65 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 146 | 175 | 153 | 163 | 809
  Male | 85 | 113 | 84 | 104 | 94 | 480
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 10 | 6 | 12 | 8 | 10 | 46
  Black | 2 | 2 | 8 | 6 | 9 | 27
  Other | 21 | 27 | 30 | 29 | 28 | 135
  White | 224 | 224 | 209 | 214 | 210 | 1081

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein (LDL-C) at Week 12
Time Frame: Baseline and 12 weeks
Population: Full Analysis Set (FAS). The FAS population includes all randomized patients with baseline (BL) value and at least one valid after-BL value. After-BL measurements up to 3 days following the last dose of double-blind study medication were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change in LDL-C
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg
Number analyzed (Participants) | 242 | 232 | 238 | 236 | 239
Percent change in LDL-C | -39.5 [-41.4 to -37.5] | -54.2 [-56.1 to -52.2] | -46.6 [-48.6 to -44.7] | -59.1 [-61.0 to -57.1] | -50.8 [-52.8 to -48.9]
Statistical Analysis 1: Comparison: Atorvastatin 10 mg vs Ezetimibe 10 mg/Simvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; ANCOVA mixed model with fixed effects for treatment, baseline LDL-C, study week, treatment by study week interaction, and a random subject effect; Mean Difference (Final Values) = -14.7, 95% CI [-17.5 to -12.0], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: Ezetimibe 10 mg/Simvastatin 20 mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.5, 95% CI [-10.3 to -4.8], Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: Ezetimibe 10 mg/Simvastatin 40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.2, 95% CI [-11.0 to -5.5], Standard Error of Mean 1.4

2. Secondary Outcome: Percentage of Patients Who Achieved LDL-C <70 mg/dL at Week 12
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent of Patients
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg
Number analyzed (Participants) | 242 | 232 | 238 | 236 | 239
Percent of Patients | 9.9 (1.92) | 51.3 (3.28) | 26.1 (2.85) | 68.2 (3.03) | 38.1 (3.14)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg vs Ezetimibe 10 mg/Simvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction. Generalized Estimating Equations (GEE); Ratio of odds = 12.62, 95% CI [7.64 to 20.83], Standard Error of Mean 3.23 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 2: Comparison: Ezetimibe 10 mg/Simvastatin 20 mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 3.83, 95% CI [2.51 to 5.85], Standard Error of Mean 0.83 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 3: Comparison: Ezetimibe 10 mg/Simvastatin 40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 3.66, 95% CI [2.39 to 5.60], Standard Error of Mean 0.79 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva

3. Secondary Outcome: Percentage of Patients Without Atherosclerosis Vascular Disease (AVD) Who Achieved LDL-C <100 mg/dL or Patients With AVD Who Achieved LDL-C <70 mg/dL at Week 12
Description: Patients with AVD Who Achieved LDL-C <70 mg/dL. AVD was defined as a history of myocardial infarction, stable angina, coronary artery procedures or evidence of clinically significant myocardial ischemia.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent of Patients
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg
Number analyzed (Participants) | 242 | 232 | 238 | 236 | 239
Percent of Patients | 45.0 (3.20) | 69.0 (3.04) | 61.3 (3.16) | 82.1 (2.50) | 69.9 (2.97)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg vs Ezetimibe 10 mg/Simvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 3.05, 95% CI [2.04 to 4.55], Standard Error of Mean 0.62 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 2: Comparison: Ezetimibe 10 mg/Simvastatin 20 mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.039, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 1.54, 95% CI [1.02 to 2.32], Standard Error of Mean 0.32 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 3: Comparison: Ezetimibe 10 mg/Simvastatin 40 mg vs Atorva 40 mg; Test type: Superiority or Other; p = 0.023, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 1.81, 95% CI [1.14 to 2.87], Standard Error of Mean 0.43 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva

4. Secondary Outcome: Percentage of Patients Who Achieved LDL-C <100 mg/dL at Week 12
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent of Patients
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg
Number analyzed (Participants) | 242 | 232 | 238 | 236 | 239
Percent of Patients | 58.7 (3.17) | 83.6 (2.43) | 76.9 (2.73) | 90.3 (1.93) | 79.5 (2.61)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg vs Ezetimibe 10 mg/Simvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 4.47, 95% CI [2.76 to 7.24], Standard Error of Mean 1.10 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 2: Comparison: Ezetimibe 10 mg/Simvastatin 20 mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.026, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 1.77, 95% CI [1.07 to 2.94], Standard Error of Mean 0.46 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 3: Comparison: Ezetimibe 10 mg/Simvastatin 40 mg vs Atorva 40 mg; Test type: Superiority or Other; p = 0.017, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 2.27, 95% CI [1.23 to 4.18], Standard Error of Mean 0.71 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva

5. Secondary Outcome: Percentage of Patients With High Risk for CHD Who Achieved LDL-C <70 mg/dL at Week 12
Description: Risk was assessed utilizing a history of established CHD or CHD risk equivalent and Framingham Risk scoring.
Time Frame: 12 Weeks
Population: Patients with High Risk for CHD in the Full Analysis Set (FAS). The FAS population includes all randomized patients with baseline (BL) value and at least one valid after-BL value. After-BL measurements up to 3 days following the last dose of double-blind study medication were included in the analysis.
Measure: Mean (Standard Error); unit: Percent of Patients
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg
Number analyzed (Participants) | 138 | 138 | 128 | 130 | 136
Percent of Patients | 10.9 (2.65) | 54.3 (4.24) | 28.9 (4.01) | 69.2 (4.05) | 38.2 (4.17)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg vs Ezetimibe 10 mg/Simvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 7.60, 95% CI [4.31 to 13.42], Standard Error of Mean 2.20 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 2: Comparison: Ezetimibe 10 mg/Simvastatin 20 mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 2.95, 95% CI [1.86 to 4.67], Standard Error of Mean 0.69 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 3: Comparison: Ezetimibe 10 mg/Simvastatin 40 mg vs Atorva 40 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 2.15, 95% CI [1.42 to 3.27], Standard Error of Mean 0.46 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva

6. Secondary Outcome: Percentage of Patients With AVD Who Achieved LDL-C <70 mg/dL at Week 12
Description: as for outcome 3
Time Frame: 12 Weeks
Population: Patients with AVD in the Full Analysis Set (FAS). The FAS population includes all randomized patients with baseline (BL) value and at least one valid after-BL value. After-BL measurements up to 3 days following the last dose of double-blind study medication were included in the analysis.
Measure: Mean (Standard Error); unit: Percent of Patients
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorva 40 mg
Number analyzed (Participants) | 70 | 81 | 79 | 79 | 72
Percent of Patients | 10.0 (3.59) | 44.4 (5.52) | 31.6 (5.23) | 65.8 (5.34) | 44.4 (5.86)
Statistical Analysis 1: Comparison: Atorvastatin 10 mg vs Ezetimibe 10 mg/Simvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 6.02, 95% CI [2.71 to 13.38], Standard Error of Mean 2.45 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 2: Comparison: Ezetimibe 10 mg/Simvastatin 20 mg vs Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.069, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 1.67, 95% CI [0.96 to 2.60], Standard Error of Mean 0.47 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva
Statistical Analysis 3: Comparison: Ezetimibe 10 mg/Simvastatin 40 mg vs Atorva 40 mg; Test type: Superiority or Other; p = 0.039, Logistic Regression using GEE — Reported p-value is multiplicity-adjusted. Hochberg procedure was used to adjust for multiple comparisons; Model include terms for treatment, baseline LDL-C, study week and treatment by study week interaction; Ratio of odds = 1.78, 95% CI 2-sided [1.10 to 2.90], Standard Error of Mean 0.44 — Ratio of odds of achieving pre-specified LDL-C level on EZ/Simva versus Atorva

ADVERSE EVENTS:
Description: AE reporting is based on number of subjects at risk. Subjects at risk are randomized subjects who received at least one dose of study drug. Five patients where excluded from the randomized population because they did not receive one dose of study drug (EZ/Simva 20 mg - 3 patients; Atorva 20 mg - 1 patient; Atorva 40 mg - 1 patient).
Groups:
- Atorvastatin 40 mg: Atorvastatin 40 mg once daily for 12 weeks
Arm/Group | Atorvastatin 10 mg | Ezetimibe 10 mg/Simvastatin 20 mg | Atorvastatin 20 mg | Ezetimibe 10 mg/Simvastatin 40 mg | Atorvastatin 40 mg
Serious Adverse Events (participants affected / at risk) | 4/257 | 8/256 | 3/258 | 3/257 | 5/256
Other Adverse Events (participants affected / at risk) | 26/257 | 32/256 | 26/258 | 32/257 | 30/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin 10 mg (N=257) | Ezetimibe 10 mg/Simvastatin 20 mg (N=256) | Atorvastatin 20 mg (N=258) | Ezetimibe 10 mg/Simvastatin 40 mg (N=257) | Atorvastatin 40 mg (N=256)
AV dissociation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mechanical complication of implant (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin 10 mg (N=257) | Ezetimibe 10 mg/Simvastatin 20 mg (N=256) | Atorvastatin 20 mg (N=258) | Ezetimibe 10 mg/Simvastatin 40 mg (N=257) | Atorvastatin 40 mg (N=256)
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 4 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 4 | 4 | 4
Nasopharyngitis (Infections and infestations) | 2 | 5 | 4 | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 4 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3 | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 2 | 3
Dizziness (Nervous system disorders) | 2 | 6 | 0 | 2 | 3
Headache (Nervous system disorders) | 1 | 5 | 3 | 3 | 2
Hypertension (Vascular disorders) | 1 | 3 | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.